CLINICAL TRIAL: NCT03316053
Title: Cell Marker Predictors in Barrett's Esophagus
Status: Active, not recruiting | Type: Observational
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1708-43
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Barrett's Esophagus Without Dysplasia
MeSH Terms: interventions — Histocompatibility Testing; Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy during endoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tissue Sample for genetic testing: Biopsy sample
  Interventions: Other: Tissue sample for genetic testing

INTERVENTIONS:
Other: Tissue sample for genetic testing — Tissue sample to be obtained during routine endoscopy

SUMMARY:
The purpose of this study is to analyze biopsied tissue samples for changes in cells and genes involved in Barrett's Esophagus.

DETAILED DESCRIPTION:
Patients with a history of Barrett's esophagus who are scheduled for a routine endoscopy will have an additional biopsy taken for genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* History of Barrett's esophagus; scheduled for routine upper endoscopy

Exclusion Criteria:

* Under 18 years of age
* Unable to consent on own behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of Barrett's esophagus
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Cell Markers | through study completion, an average of 1 year
  Identify genes involved in Barrett's Esophagus

CONTACTS AND LOCATIONS:
Overall Officials: Michael Georgetson, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- The Guthrie Clinic, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No